CLINICAL TRIAL: NCT06251869
Title: Electrocoagulation vs. Cold Knife Cutting in Joint Arthroplasty: A Comparative Analysis in Knee and Hip Replacement
Brief Title: Electrocoagulation vs. Cold Knife Cutting in Joint Arthroplasty (Electrocoagulation vs Scalpel)
Acronym: evs
Status: Recruiting | Type: Observational
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Benea Horea, Assoc. Professor, Orthopedics and Traumatology Surgeon, MD, PhD, Iuliu Hatieganu University of Medicine and Pharmacy
Other Study IDs: umfcj002
Record Dates: First submitted 2023-12-14; First posted 2024-02-09 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Compassion
Keywords: electrocoagulation; cold knife; scalpel; joint arthroplasty; knee replacement; hip replacement; comparative analysis; surgical techniques; orthopedics; outcome assessment
MeSH Terms: conditions — Hyperthermia | interventions — Arthroplasty, Replacement, Hip; Electrocoagulation; Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- hip electrocoagulation: group subjected to the use of electrocoagulation
  Interventions: Procedure: total hip arthroplasty with electrocoagulation
- hip scalpel: group subjected to the use of traditional hemostatic technique
  Interventions: Procedure: total hip arthroplasty without electrocoagulation
- knee electrocoagulation: group subjected to the use of electrocoagulation
  Interventions: Procedure: total knee arthroplasty with electrocoagulation
- knee scalpel: group subjected to the use of traditional hemostatic technique
  Interventions: Procedure: total knee arthroplasty without electrocoagulation

INTERVENTIONS:
Procedure: total hip arthroplasty with electrocoagulation — using normal technique
  Groups: hip electrocoagulation
Procedure: total hip arthroplasty without electrocoagulation — using only scalpel and pean as hemostasis and incision
  Groups: hip scalpel
Procedure: total knee arthroplasty with electrocoagulation — using normal technique
  Groups: knee electrocoagulation
Procedure: total knee arthroplasty without electrocoagulation — using only scalpel and pean as hemostasis and incision
  Groups: knee scalpel

SUMMARY:
Comparison of clinical outcomes of electrocoagulation and non-electrocoagulation techniques in total hip and knee arthroplasty surgery

DETAILED DESCRIPTION:
Objectives:

A. To evaluate the effectiveness of electrocoagulation:

* To measure the reduction in intraoperative bleeding volume when using electrocoagulation.
* Analyse the impact of electrocoagulation on surgical visibility and accuracy during implant placement.

B. Comparison of surgical outcomes:

* Investigate the incidence of intra- and postoperative complications, such as incidental vascular-nerve injury, wound infections, deep vein thrombosis, and implant-related problems, in patients operated on with electrocoagulation versus techniques without electrocoagulation.
* Examine the influence of haemostatic technique on the need for blood transfusion during or after surgery.
* Evaluation of long-term functional outcomes and patient satisfaction, including joint stability and range of motion, in both groups.

C. Review of patient recovery and period of hospitalization:

* Analysis of the impact of electrocoagulation on length of hospitalisation, and time to ambulation.
* Assessment of postoperative pain levels and analgesic medication use between the two groups.
* Patients' return to daily activities and overall quality of life after surgery.

D. Comparison of data obtained with other studies conducted internationally.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given informed consent to the procedure
* Patients admitted over 18 years of age
* Patients with pathology requiring primary joint replacement (symptomatic gonarthrosis/coxarthrosis, Avascular necrosis (AVN) of the femoral head , femoral neck fractures, etc)

Exclusion Criteria:

* Contraindications for major surgery or anaesthesia
* Patients with active infections that could interfere with outcome assessment
* Patients unable to give informed consent for psychological or cognitive reasons
* Severe medical conditions such as coagulopathies that may significantly influence outcomes
* Patients unable or unwilling to adhere to the required follow-up period
* Patients who died during the study period
* Patients with revision prosthesis operations

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: anyone who needs a hip/knee replacemnt
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) knee subjective score | the test will be administered pre operation, 2 weeks post-operation, 6 weeks post-op, 3 months post-op, 6 months post-op, 1 year post-op
  to objectify the recovery, score is on a scale, higher values mean a worse outcome, scale 0-168
Western Ontario and McMaster Universities Osteoarthritis index (WOMAC) subjective score | the test will be administered pre operation, 2 weeks post-operation, 6 weeks post-op, 3 months post-op, 6 months post-op, 1 year post-op
  to objectify the recovery, score is on a scale, higher values mean a worse outcome, scale 0-96 .
International Knee Documentation Committee (IKDC) objective form | the test will be administered pre operation, 2 weeks post-operation, 6 weeks post-op, 3 months post-op, 6 months post-op, 1 year post-op
  to objectify the recovery, score has different classifications on a scale from A to D, the latter being the worse outcome .
Harris Hip Score | the test will be administered pre operation, 2 weeks post-operation, 6 weeks post-op, 3 months post-op, 6 months post-op, 1 year post-op
  to objectify the recovery, score is on a scale, higher values mean a better outcome, scale 0-100 .
Hip dysfunction and Osteoarthritis Outcome Score for Joint Replacement (HOOS-JR) hip subjective score | the test will be administered pre operation, 2 weeks post-operation, 6 weeks post-op, 3 months post-op, 6 months post-op, 1 year post-op
  to objectify the recovery, score is on a scale, higher values mean a worse outcome, scale 0-24 .
Forgotten Joint Score | the test will be administered 2 weeks post-operation, 6 weeks post-op, 3 months post-op, 6 months post-op, 1 year post-op
  to objectify the recovery, score is on a scale, higher values mean a worse outcome, scale 0-48 .

SECONDARY OUTCOMES:
hemaglobin levels | the hemaglobin levels will be registered pre-operation, then post-op day: 1, 2, 3, 4, and 5. Then at 2 weeks post-operation, 6 weeks, and 3 months
  for blood loss objectification .
leucocyte levels | the leucocyte levels will be registered pre-operation, then post-op day: 1, 2, 3, 4, and 5. Then at 2 weeks post-operation, 6 weeks, and 3 months
  for infection objectification .
thrombocyte levels | the thrombocyte levels will be registered pre-operation, then post-op day: 1, 2, 3, 4, and 5. Then at 2 weeks post-operation, 6 weeks, and 3 months
  for blood loss objectification .
mobilisation intervals of the patient | through hospital stay of patient approximatively 4-7 days
  the investigators will asses the time for the self-mobilisation of the patient to sit at the bed's edge, and then mobilisation with a walking aid like a walking frame. .
joint hyperextension angle | the measurements will be registered pre-operative, then 2 weeks post-operation, 6 weeks post-op, 3 months post-op, 6 months post-op, 1 year post-op
  to objectify the recovery, the measurement will be done with a measuring angle during objective evaluation. .
joint flexion angle | the measurements will be registered pre-operative, then 2 weeks post-operation, 6 weeks post-op, 3 months post-op, 6 months post-op, 1 year post-op
  to objectify the recovery, the measurement will be done with a measuring angle during objective evaluation. .
genu flexum angle | the measurements will be registered pre-operative, then 2 weeks post-operation, 6 weeks post-op, 3 months post-op, 6 months post-op, 1 year post-op
  to objectify the recovery, the measurement will be done with a measuring angle during objective evaluation. .
joint external rotation angle | the measurements will be registered pre-operative, then 2 weeks post-operation, 6 weeks post-op, 3 months post-op, 6 months post-op, 1 year post-op
  to objectify the recovery, the measurement will be done with a measuring angle during objective evaluation. .
joint internal rotation angle | the measurements will be registered pre-operative, then 2 weeks post-operation, 6 weeks post-op, 3 months post-op, 6 months post-op, 1 year post-op
  to objectify the recovery, the measurement will be done with a measuring angle during objective evaluation. .
joint abduction angle | the measurements will be registered pre-operative, then 2 weeks post-operation, 6 weeks post-op, 3 months post-op, 6 months post-op, 1 year post-op
  to objectify the recovery, the measurement will be done with a measuring angle during objective evaluation. .
joint adduction angle | the measurements will be registered pre-operative, then 2 weeks post-operation, 6 weeks post-op, 3 months post-op, 6 months post-op, 1 year post-op
  to objectify the recovery, the measurement will be done with a measuring angle during objective evaluation. .
Number of participants with complications | through study completion, an average of 1 year
  to objectify the superiority of one technique over the other, higher number signifies a worse outcome .

CONTACTS AND LOCATIONS:
Overall Officials: Benea R Horea, MD, Principal Investigator — Iuliu Hatieganu University of Medicine and Pharmacy, Cluj-Napoca, Romania
Locations (1):
- Clinica Ortopedie-Traumatologie, Secția 2, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sonntag R, Gibmeier J, Pulvermacher S, Mueller U, Eckert J, Braun S, Reichkendler M, Kretzer JP. Electrocautery Damage Can Reduce Implant Fatigue Strength: Cases and in Vitro Investigation. J Bone Joint Surg Am. 2019 May 15;101(10):868-878. doi: 10.2106/JBJS.18.00259. PMID 31094978
- [Background] Lacitignola L, Desantis S, Izzo G, Staffieri F, Rossi R, Resta L, Crovace A. Comparative Morphological Effects of Cold-Blade, Electrosurgical, and Plasma Scalpels on Dog Skin. Vet Sci. 2020 Jan 12;7(1):8. doi: 10.3390/vetsci7010008. PMID 31940962
- [Background] Lin W, Dai Y, Niu J, Yang G, Li M, Wang F. Scalpel can achieve better clinical outcomes compared with electric cautery in primary total knee arthroplasty: a comparison study. BMC Musculoskelet Disord. 2020 Jun 29;21(1):409. doi: 10.1186/s12891-020-03457-1. PMID 32600294
- [Background] Behrend H, Giesinger K, Giesinger JM, Kuster MS. The "forgotten joint" as the ultimate goal in joint arthroplasty: validation of a new patient-reported outcome measure. J Arthroplasty. 2012 Mar;27(3):430-436.e1. doi: 10.1016/j.arth.2011.06.035. Epub 2011 Oct 13. PMID 22000572
- [Background] Cadeddu JA. Re: Lateral temperature spread of monopolar, bipolar and ultrasonic instruments for robot-assisted laparoscopic surgery. J Urol. 2015 Jan;193(1):129. doi: 10.1016/j.juro.2014.10.014. Epub 2014 Oct 12. No abstract available. PMID 25523661
- [Background] Tammachote N, Kanitnate S. Electric cautery does not reduce blood loss in primary total knee arthroplasty compared with scalpel only surgery a double-blinded randomized controlled trial. Int Orthop. 2018 Dec;42(12):2755-2760. doi: 10.1007/s00264-018-4048-y. Epub 2018 Jul 3. PMID 29968137
- [Background] Ozturk K, Kaya I, Turhal G, Ozturk A, Gursan G, Akyildiz S. A comparison of electrothermal bipolar vessel sealing system and electrocautery in selective neck dissection. Eur Arch Otorhinolaryngol. 2016 Nov;273(11):3835-3838. doi: 10.1007/s00405-016-3999-0. Epub 2016 Mar 23. PMID 27007131
- [Background] Groot G, Chappell EW. Electrocautery used to create incisions does not increase wound infection rates. Am J Surg. 1994 Jun;167(6):601-3. doi: 10.1016/0002-9610(94)90106-6. PMID 8209936